CLINICAL TRIAL: NCT02995265
Title: Use of a Robotic Exoskeleton to Promote Walking Recovery After Stroke - Phase 2
Brief Title: Exoskeleton for Post-Stroke Recovery of Ambulation
Acronym: ExStRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Janice Eng, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H15-01339
Record Dates: First submitted 2016-12-07; First posted 2016-12-16 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Conditions
Keywords: Exoskeleton; Stroke; Walking; Rehabilitation
MeSH Terms: conditions — Disease; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Exoskeleton Program (Experimental): Exoskeleton-based walking rehabilitation until discharge (or to a maximum of 8 weeks), 3 - 5 days a week for 30-60 minutes per session. Participants will be assessed upon admission to the study, discharge, as well as at 6 months post-stroke. The exoskeleton will allow standing and walking with full weight bearing from the first sessions in rehabilitation.
  Interventions: Device: Exoskeleton Program
- Usual Care Program (Active Comparator): Standard physiotherapy stroke rehabilitation which includes training for regaining walking as well as other functional tasks, 3 - 5 days a week for 30-60 minutes per session until discharge (or to a maximum of 8 weeks). Participants will be assessed upon admission to the study, discharge, as well as at 6 months post-stroke.
  Interventions: Other: Usual Care Program

INTERVENTIONS:
Device: Exoskeleton Program — Subjects will wear the exoskeleton device at each physiotherapy session to work on improving mobility and walking ability.
  Arms: Exoskeleton Program
Other: Usual Care Program — Subjects will receive hands-on physiotherapy to improve their mobility and walking ability. Physiotherapy session will be tailored to subject individually by their therapist.
  Arms: Usual Care Program

SUMMARY:
To determine the effect of using a robotic exoskeleton to allow walking practice after stroke, compared to usual physiotherapy care, on recovery of walking ability and secondary outcomes.

DETAILED DESCRIPTION:
Participants admitted to inpatient stroke rehabilitation for physiotherapy services will be randomly assigned to either the Exoskeleton Program or Usual Care Program.

Individuals in the Exoskeleton Program will have their usual physiotherapy sessions replaced with the exoskeleton intervention. The exoskeleton will allow standing and walking from the first sessions in rehabilitation, as the exoskeleton provides the physical support to allow walking in full weight-bearing without being limited by therapist fatigue and lifting requirements. Individuals in the Usual Care Program will receive standard physiotherapy care, which is individualized and hands-on with their therapist to regain walking, mobility, and independent function.

Both groups will be conducted 3-5 days a week, 30-60 minutes per session until discharge (to a maximum of 8 weeks). Participants will be assessed at baseline, discharge, and 6-months after starting rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Have been admitted to a hospital unit for stroke treatment
* Stroke within last 3 months
* One-sided hemiparesis
* 19 years or older
* Requires 2-person assist to walk
* Able to communicate and follow instructions
* Prescribed to receive physiotherapy care

Exclusion Criteria:

* Stroke of non-vascular origin (e.g. tumour, infection)
* Significant musculoskeletal or other neurological condition
* Co-morbidities that would preclude activity
* Pregnant
* Unable to walk prior to stroke
* <60 inches or >74 inches in height
* >220 pounds in weight
* Joint contractures or spasticity that would limit safe use of the Ekso exoskeleton

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-02-08 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Walking ability - Functional Ambulation Category | Rehabilitation Discharge (generally 4-6 weeks, up to 8 weeks)

SECONDARY OUTCOMES:
5-Metre Walk Test (5MWT) | Discharge (generally 4-6 weeks, up to 8 weeks), 6 months from admission
6-Minute Walk Test (6MWT) | Discharge (generally 4-6 weeks, up to 8 weeks), 6 months from admission
Berg Balance Scale (BBS) | Discharge (generally 4-6 weeks, up to 8 weeks), 6 months from admission
Health-related Quality of Life (SF-36) | Discharge (generally 4-6 weeks, up to 8 weeks), 6 months from admission
Depressive Symptoms (PHQ-9) | Discharge (generally 4-6 weeks, up to 8 weeks), 6 months from admission
Days to independent walking | Discharge (generally 4-6 weeks, up to 8 weeks)
  The number of days from admission until the participant is able to walk without any manual assistance from a therapist will be recorded.
Motor impairment/recovery of the lower extremity (Fugl-Meyer Lower) | Discharge (generally 4-6 weeks, up to 8 weeks), 6 months from admission
Cognition - Montreal Cognitive Assessment (MoCA) | Discharge (generally 4-6 weeks, up to 8 weeks), 6 months from admission
Functional Ambulation Category | 6 Months from admission
Daily step count | 6 months from admission
  ActivPAL recording over 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Janice J Eng, PhD, Principal Investigator — Department of Physical Therapy, University of British Columbia
Locations (3):
- Canada (3):
  - Glenrose Rehabilitation hospital, Edmonton, Alberta
  - GF Strong Rehab Centre, Vancouver, British Columbia
  - Parkwood Institute, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Louie DR, Mortenson WB, Lui M, Durocher M, Teasell R, Yao J, Eng JJ. Patients' and therapists' experience and perception of exoskeleton-based physiotherapy during subacute stroke rehabilitation: a qualitative analysis. Disabil Rehabil. 2022 Dec;44(24):7390-7398. doi: 10.1080/09638288.2021.1989503. Epub 2021 Oct 25. PMID 34694189
- [Derived] Louie DR, Mortenson WB, Durocher M, Schneeberg A, Teasell R, Yao J, Eng JJ. Efficacy of an exoskeleton-based physical therapy program for non-ambulatory patients during subacute stroke rehabilitation: a randomized controlled trial. J Neuroeng Rehabil. 2021 Oct 10;18(1):149. doi: 10.1186/s12984-021-00942-z. PMID 34629104
- [Derived] Louie DR, Mortenson WB, Durocher M, Teasell R, Yao J, Eng JJ. Exoskeleton for post-stroke recovery of ambulation (ExStRA): study protocol for a mixed-methods study investigating the efficacy and acceptance of an exoskeleton-based physical therapy program during stroke inpatient rehabilitation. BMC Neurol. 2020 Jan 28;20(1):35. doi: 10.1186/s12883-020-1617-7. PMID 31992219